CLINICAL TRIAL: NCT04086173
Title: Effects of Probiotic Treatment on Body Composition and Insulin Resistance in Patients With Obesity Grade II and III and Its Association With Changes in Intestinal Microbiota
Brief Title: Probiotics on Body Composition and Insulin Resistance in Patients With Obesity and Its Association With Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Collaborators: Italmex Pharma (Unknown); Medix Farma (Unknown); National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Nayely Garibay Nieto, Head Child and Adolescent Obesity Clinic, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00000
Record Dates: First submitted 2019-03-05; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Obesity; Insulin Resistance; Microbial Colonization
MeSH Terms: conditions — Obesity; Insulin Resistance; Communicable Diseases | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized placebo-controlled clinical assay
Who Masked: Participant, Care Provider
Masking Description: Neither the participant nor the Care provider administrating treatment will know the type of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Subjects will be randomly assigned to receive a daily nightly dose (4 capsules) of probiotics for 16 weeks. Probiotics (LACTIPAN®) include 2.5 billion CFU of 6 different strains of live microorganisms, such as Lactobacillus acidophilus (1.0 x 109 CFU), Lactobacillus casei (1.0 x 109 CFU), Lactobacillus rhamnosus (4.4 x 108 CFU), Lactobacillus plantarum (1.76 x 108 CFU), Bifidobacterium infantis (2.76 x 107 CFU), Streptococcus thermophilus (6.66 x 105 CFU) and 50 mg of oligofructose enriched inulin.
  Interventions: Dietary Supplement: Probiotics
- Control group (Placebo Comparator): Subjects will be randomly assigned to receive a daily nightly dose (4 capsules) of placebo for 16 weeks. Placebo presentation will have the same aspect as those of the probiotic treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics will be administered at night and will consist of 4 capsules
  Arms: Study group
Other: Placebo — Placebo
  Arms: Control group

SUMMARY:
This study aims to evaluate the modifications in body composition and insulin resistance state in patients with grade II and III obesity included in an interventional lifestyle changes program and treated with probiotics (1 x 1011 CFU) or placebo for 16 weeks and its associations with intestinal microbiota behaviour

DETAILED DESCRIPTION:
A randomized placebo-controlled clinical trial will take place in which both arms will be included in an interventional lifestyle changes program at the Clinic for Integral Treatment of patients with Diabetes and Obesity. The study group will be treated with probiotics (1 x 1011 CFU) for 16 weeks and will be compared to a control group who will receive placebo.

Changes in body composition (weight, BMI, fat percentage, fat mass, lean body mass) and insulin resistance indexes (HOMA, insulin sensitivity index and Quicki) will be evaluated in patients with obesity receiving probiotics (1 x 1011 CFU) for 16 weeks, and compared to a placebo group.

Changes in metabolic profile (glucose tolerance test, glycosylated haemoglobin, lipid profile, leptin and transaminases) in patients with obesity receiving probiotics (1 x 1011 CFU) for 16 weeks, and compared to a placebo group.

Changes in microRNAs profile (miR-133 and miR-27 in patients with obesity receiving probiotics (1 x 1011 CFU) for 16 weeks, and compared to a placebo group.

The threshold for basic tastes will be evaluated (salted, bitter, acid, sweet) and will be evaluated in those patients receiving probiotics (1 x 1011 CFU) for 16 weeks, and compared to the group receiving only placebo.

Changes in intestinal microbiota behaviour will be evaluated in participants with obesity receiving probiotics (1 x 1011 CFU) for 16 weeks, and compared to the group receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade II y III obesity (IMC > or = 35 Kg/m2), who receive the initial evaluation at the Integral Attention Clinic for Diabetes and Obesity at Hospital General de México
* Patients who signed informed consent.

Exclusion Criteria:

* Diabetes mellitus 2
* Secondary causes of obesity (hypothyroidism, Cushing syndrome).
* Patients receiving pharmacological treatment that may affect lipid or glucose metabolism.
* Patients who received broad-spectrum antibiotics during the 4 previous weeks.
* Ingestion of products that contain probiotics.
* Relevant changes in diet habits during the 4 previous weeks
* Intestinal Malabsorption disorders ( inflammatory bowel disease, chronic diarrhea, C. difficile infection).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in fat mass in patients with obesity | 16 weeks
  Evaluate changes in fat mass kilograms after probiotics treatment in patients with obesity, by bioelectrical impedance analysis
Changes in fat percentage in patients with obesity | 16 weeks
  Evaluate changes in fat percentage after probiotics treatment in patients with obesity, by bioelectrical impedance analysis
Changes in body mass index in patients with obesity | 16 weeks
  Evaluate changes in body mass index after probiotics treatment in patients with obesity. Calculated with the weight in kilograms divided by the square of the height in meters
Changes in weight in patients with obesity | 16 weeks
  Evaluate changes in weight kilograms after probiotics treatment in patients with obesity
Changes in lean body mass in patients with obesity | 16 weeks
  Evaluate changes in lean body mass kilograms after probiotics treatment in patients with obesity, by bioelectrical impedance analysis
Changes in Insulin resistance indexes | 16 weeks
  Modification in HOMA index after probiotics treatment in patients with obesity
Changes in Insulin sensitivity indexes | 16 weeks
  Modification in insulin sensitivity index after probiotics treatment in patients with obesity
Changes in Quicki insulin sensitivity index | 16 weeks
  Modification in Quicki index after probiotics treatment in patients with obesity

SECONDARY OUTCOMES:
Changes in glucose tolerance test | 16 weeks
  Evaluate changes in glucose tolerance test after treatment with probiotics in patients with obesity. By using plasma concentrations of insulin and glucose obtained during 120 min of a standard (75 g glucose).
Changes in glycated haemoglobin | 16 weeks
  Evaluate changes in percentage glycated haemoglobin after treatment with probiotics in patients with obesity. Obtain by capillary electrophoresis system
Changes in triglycerides | 16 weeks
  Evaluate changes in triglycerides (mg/dL) after treatment with probiotics in patients with obesity
Changes in total cholesterol | 16 weeks
  Evaluate changes in total cholesterol (mg/dL) after treatment with probiotics in patients with obesity
Changes in HDL cholesterol | 16 weeks
  Evaluate changes in HDL cholesterol (mg/dL) after treatment with probiotics in patients with obesity
Changes in LDL cholesterol | 16 weeks
  Evaluate changes in LDL cholesterol (mg/dL) after treatment with probiotics in patients with obesity
Changes in uric acid | 16 weeks
  Evaluate changes in uric acid (mg/dL) after treatment with probiotics in patients with obesity
Changes in aspartate aminotransferase | 16 weeks
  Evaluate changes in aspartate aminotransferase (U/L) after treatment with probiotics in patients with obesity
Changes in alanine aminotransferase | 16 weeks
  Evaluate changes in alanine aminotransferase (U/L) after treatment with probiotics in patients with obesity
Changes in leptin | 16 weeks
  Evaluate changes in leptin (ng/mL) after treatment with probiotics in patients with obesity

OTHER OUTCOMES:
Changes in microRNAs | 16 weeks
  Evaluate changes in miR-133 and miR-27 after treatment with probiotics in patients with obesity
Compare threshold for basic tastes | 16 weeks
  Evaluate differences in basic taste thresholds (sour, salty, sweet and bitter) after treatment with probiotics in patients with obesity
Changes in intestinal microbiota | 16 weeks
  Evaluate differences in intestinal microbiota behaviour after treatment with probiotics in patients with obesity

CONTACTS AND LOCATIONS:
Overall Officials: Nayely Garibay-Nieto, MSc, Principal Investigator — Hospital General de Mexico Eduardo Liceaga
Locations (1):
- Hospital General de México "Dr. Eduardo Liceaga", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banegas JR, Lopez-Garcia E, Gutierrez-Fisac JL, Guallar-Castillon P, Rodriguez-Artalejo F. A simple estimate of mortality attributable to excess weight in the European Union. Eur J Clin Nutr. 2003 Feb;57(2):201-8. doi: 10.1038/sj.ejcn.1601538. PMID 12571650
- [Background] Neish AS. Microbes in gastrointestinal health and disease. Gastroenterology. 2009 Jan;136(1):65-80. doi: 10.1053/j.gastro.2008.10.080. Epub 2008 Nov 19. PMID 19026645
- [Background] Hooper LV, Wong MH, Thelin A, Hansson L, Falk PG, Gordon JI. Molecular analysis of commensal host-microbial relationships in the intestine. Science. 2001 Feb 2;291(5505):881-4. doi: 10.1126/science.291.5505.881. PMID 11157169
- [Background] Jalanka J, Mattila E, Jouhten H, Hartman J, de Vos WM, Arkkila P, Satokari R. Long-term effects on luminal and mucosal microbiota and commonly acquired taxa in faecal microbiota transplantation for recurrent Clostridium difficile infection. BMC Med. 2016 Oct 11;14(1):155. doi: 10.1186/s12916-016-0698-z. PMID 27724956
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309